CLINICAL TRIAL: NCT00138489
Title: Protocol 3B Susceptibility to Plasmodium Vivax Infection and Malaria During Early Childhood
Brief Title: Papua New Guinean Duffy Negativity And Vivax Malar
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 02-004; Protocol 3B
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2007-10

CONDITIONS: Plasmodium Vivax Malaria
Keywords: Malaria, Papua New Guinea, infants, children
MeSH Terms: conditions — Malaria, Vivax; Malaria

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to learn more about vivax malaria in very young children, how the growth of children is affected by malaria infections, and how inherited traits protect children from getting malaria. Participants will be 266 children 24 months of age or younger who live in certain villages in East Sepik Province, Papua New Guinea, where malaria is very common. The study also will find out how malaria spreads in the area. By learning how and when a child develops resistance to vivax malaria, researchers can try to find ways to help people from getting it. And, they can get a better understanding of how inherited traits influence all types of malaria infections. In this study, the parent and child will be visited by the study team or health workers every week to check health and bednet use. Every 2 weeks, the study team will take a small blood sample to check for malaria and take measurements to study the child's growth. Participants will be followed for up to 2 years.

DETAILED DESCRIPTION:
This study specifically seeks to document infection by Plasmodium species parasites in a prospective longitudinal study using blood smear and polymerase chain reaction (PCR)/Ligase Detection Reaction (LDR) diagnostic techniques and to determine when a child becomes susceptible to blood-stage malaria in a cohort of non-immune children from villages where a genetic polymorphism that blocks expression of Duffy (Fy) blood group antigen has been identified. The goal of this project is to prospectively study the natural history of Plasmodium vivax malaria in a malaria-endemic region of Papua New Guinea among a cohort of children 24 months of age and older for a period of up to two years. The primary objectives of this study are to: 1) determine the mean time to first P. vivax infection, and 2) determine the incidence rate of P. vivax infection. The secondary objectives of this study are to: 1) assess the impact of recurrent Plasmodium infections on child growth, 2) estimate the sensitivity and specificity of blood smear versus PCR-based diagnostic methods for P. vivax infection, and 3) evaluate the effect of the FY genotype on P. vivax malaria. Cross-sectional malaria prevalence data based on blood smear diagnosis suggest that the risk of malaria is extremely low during infancy in this population. Therefore, at the start of the study, children 12 months of age and younger will be eligible for the study, and all new births occurring over the next 15 months will be added to the cohort ensuring that the last newborn will have a minimum of 9 months of follow-up. All children enrolled in this study will be followed weekly to detect clinical malaria and biweekly blood samples will be taken for the detection of asymptomatic malaria. Follow-up will continue for a period of up to 2 years until participants reach 24 months of age, or withdraw from the study or until the study ends, whichever event comes first.

ELIGIBILITY:
Inclusion Criteria:

The following criteria are applicable to this study. All three of the inclusion criteria must be met.

< = 12 months of age at the time of eligibility assessment Residence in a designated study village Parental / legal guardian consent

Participants who move outside the study area during the course of the study will be dropped from further participation. However, data collected to that point may be included in statistical analyses. Parental consent to study is essential. No blood samples or measurements will be taken on a child without informed consent.

Exclusion Criteria:

The following exclusion criteria are applicable to this study. Any one or more of the criteria is sufficient to exclude study participation.

> 12 months of age at the time of eligibility assessment Chronic illness, severe malnutrition, permanent disability, or a congenital malformation that prevents or impedes study participation Short-term, temporary residence (less than 6 months) in a designated study village Residence in a village outside of the study area Parental refusal to consent to study

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 266
Dates: Start 2004-02-10

CONTACTS AND LOCATIONS:
Locations (1):
- Papua New Guinea Institute of Medical Research, Goroka, Papua New Guinea